CLINICAL TRIAL: NCT02690909
Title: A Prospective, Post-marketing, Single-arm, Open Label, Multi-center Clinical Study to Evaluate the Safety and Efficacy of the ReDy™ Renal Denervation System in the Treatment of Patients With Uncontrolled Hypertension
Brief Title: A Study to Evaluate Safety and Efficacy of the Redy™ Renal Denervation System in the Treatment of Patients With Uncontrolled Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renal Dynamics GmbH (Industry)
Collaborators: Biosensors Europe SA (Industry); Physio-Logic Ltd. Israel (Unknown); AmeRuss Clinical Trials LLC, USA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD1501
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension Resistant to Conventional Therapy
Keywords: Uncontrolled Hypertension; Resistant Hypertension; Renal Denervation
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Redy™ Renal Denervation System (Experimental): Renal Denervation System
  Interventions: Device: Redy™ Renal Denervation System

INTERVENTIONS:
Device: Redy™ Renal Denervation System — Renal Denervation System

SUMMARY:
The ReDy™ System (Renal Dynamics) is a renal denervation device incorporating a variety of ablation features and technical improvements over previously designed systems into a single product. It is intended to treat uncontrolled (drug-resistant) hypertension by RF ablation of the sympathetic nerve network surrounding the renal arteries.

This study will be carried out to validate the safety and the efficacy of the ReDy™ Renal Denervation device and to demonstrate that it performs according to its intended use, i.e. the treatment of patients with uncontrolled hypertension.

ELIGIBILITY:
Inclusion criteria:

1. Patient has established hypertension (diagnosed ≥12 months prior to screening) and is on a guideline based stable drug regimen (≥ 4 weeks), consisting of ≥3 anti-hypertensive medications of different classes including a diuretic;
2. Office systolic blood pressure >150 mmHg;
3. Patient has (under directly observed therapy) average daytime systolic blood pressure values > 140 mmHg by 24h ambulatory blood pressure monitoring;
4. Patient is ≥ 18 and ≤ 75 years of age at time of consent;
5. Patient must be able and willing to comply with the required follow-up schedule;
6. Patient must be able and willing to provide written informed consent;

Exclusion criteria:

1. Patient has known significant reno-vascular abnormalities such as renal artery stenosis > 30%;
2. Patient has "Isolated Systolic Hypertension" with a diastolic blood pressure < 90 mmHg;
3. Evidence or history of secondary hypertension, other than sleep apnea syndrome;
4. Patient has a history of prior renal angioplasty, renal denervation, indwelling renal stents, and/or abdominal aortic stent graft placement;
5. Patient has significant valvular heart disease;
6. Patient has known coagulation abnormalities;
7. Patient life expectancy is < 12 months, as estimated by the study Investigator;
8. Patient is participating in another clinical study, which is before its primary endpoint and/or has the potential to impact his/her hypertension management (pharmaceutical / device);
9. Patient is pregnant, nursing, or of childbearing potential and is not using adequate contraceptive methods;
10. Patient has active systemic infection;
11. Patient has small <4.0 mm in diameter, large >6.5 mm in diameter or short <20.0 mm in length, multiple main, or highly tortuous renal arteries;
12. Patient has impaired renal function with an estimated GFR <45 mL/min per 1.73 m2 using the Modification of Diet in Renal Disease (MDRD) formula;
13. Patient had a renal transplant or is awaiting a renal transplant;
14. Patient has a known intolerance for x-ray contrast agent that cannot be adequately controlled with pre-medication;
15. Any medical condition as estimated by the Study Investigator that may harm patient or jeopardize study participation, the interpretation of study results or may impede the ability to obtain informed consent (e.g., mental condition);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Device-related adverse events at 1-month follow-up post treatment | 1-month post treatment
  Incidence of device-related Adverse Events at 1-month follow-up post treatment

SECONDARY OUTCOMES:
Peri-procedural Adverse Events at 1-month follow-up post treatment | 1-month post treatment
  Incidence of peri-procedural Adverse Events at 1-month follow-up post treatment
Device-related Adverse Events at 3 and 6 months follow-up post treatment | 3 and 6 months post treatment
  Incidence of device-related Adverse Events at 3 and 6 months follow-up post treatment
Reduction of average systolic daytime blood pressure assessed by 24h ABPM at 3-months | 3 months post treatment
  Reduction of average systolic daytime blood pressure as assessed by 24h ambulatory blood pressure monitoring at 3-month compared to baseline
Reduction of office systolic blood pressure at 1, 3 and 6 months post treatment | 1, 3 and 6 months post treatment
  Reduction of office systolic blood pressure at 1, 3 and 6 months post treatment
Reduction of office diastolic blood pressure at 1, 3 and 6 months post treatment | 1, 3 and 6 months post treatment
  Reduction of office diastolic blood pressure at 1, 3 and 6 months post treatment
Blood pressure control to guideline recommended target blood pressure values at 1, 3 and 6 months post treatment | 1, 3 and 6 months post treatment
  Blood pressure control to guideline recommended target blood pressure values at 1, 3 and 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Felix Mahfoud, MD, Principal Investigator — Saarland University Medical Center Homburg, Germany
Locations (10):
- Belgium (2):
  - OLV Onze-Lieve-Vrouwziekenhuis, Aalst
  - ZNA Middelheim Hospital, Antwerp
- Germany (2):
  - Asklepios Klinik St. Georg, Hamburg
  - Saarland University Medical Center, Homburg
- Semmelweis University, Budapest, Hungary
- Galway University Hospital, Galway, Ireland
- Kaplan Medical Center, Rehovot, Israel
- The Cardinal Stefan Wyszyński Institute of Cardiology, Warsaw, Poland
- Academician E.N. Meshalkin Novosibirsk State Research Institute of Circulation Pathology, Novosibirsk, Russia
- KCS Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No